CLINICAL TRIAL: NCT01652872
Title: Strategies Using Darbepoetin Alfa to Avoid Transfusions in Chronic Kidney Disease
Acronym: START-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110226
Record Dates: First submitted 2012-06-07; First posted 2012-07-30 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Anemia in Chronic Kidney Disease Patients Not on Dialysis
Keywords: anemia; chronic kidney disease; kidney disease; renal failure
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Diseases; Renal Insufficiency | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hb-Based Titration Group (Active Comparator): Participants received darbepoetin alfa as a subcutaneous (SC) injection once every 4 weeks (Q4W) for up to 96 weeks. The dose of darbepoetin alfa was titrated based on the Hb concentration on the date of the visit, the corresponding Hb rate of rise (ROR), and the previously assigned dose. Doses were reduced if Hb exceeded 10.5 g/dL or Hb ROR exceeded 1.0 g/dL/4W. When darbepoetin alfa therapy was withheld per the dosing algorithm, placebo was administered. The starting dose of darbepoetin alfa was 0.45 micrograms/kilogram (mcg/kg) and the protocol specified doses ranged from 10 to 300 mcg.
  Interventions: Biological: Darbepoetin alfa; Other: Placebo
- Fixed Dose Group (Experimental): Participants received darbepoetin alfa as a SC injection Q4W at the same dose as assigned at the time of randomization for the duration of the 96 week treatment period. There was 1 exception to the fixed dose strategy: if the Hb was > 12.0 g/dL, darbepoetin alfa therapy was withheld and placebo administered. Once the Hb fell to < 10.0 g/dL, darbepoetin alfa therapy resumed at the same dose. The starting dose of darbepoetin alfa was 0.45 mcg/kg and the protocol specified doses ranged from 10 to 300 mcg.
  Interventions: Biological: Darbepoetin alfa; Other: Placebo

INTERVENTIONS:
Biological: Darbepoetin alfa — Darbepoetin alfa was presented as single use prefilled syringes (PFS). Investigational product was administered SC Q4W for the duration of the treatment period.
  Other Names: Aranesp
Other: Placebo — Placebo was presented as single use PFS. Participants received a SC placebo injection in place of darbepoetin alfa therapy when the dose of study drug was withheld per the dosing algorithm for the duration of the treatment period.

SUMMARY:
A phase 3, multicenter, randomized, double-blind, parallel group study. Anemic subjects with chronic kidney disease (CKD) and not on dialysis will be randomized 1:1 to 1 of 2 dosing strategies to evaluate the proportion of subjects receiving at least one red blood cell (RBC) transfusion. In the haemoglobin (Hb)-based titration group, darbepoetin alfa doses will be titrated to maintain Hb ≥ 10.0 grams/deciliter (g/dL). In the fixed dose group, subjects will receive a fixed dose of darbepoetin alfa. Treatment group, darbepoetin alfa doses, and protocol specified Hb concentrations will be blinded. Subjects will be followed for approximately 2 years from the date of randomization.

DETAILED DESCRIPTION:
The study is a phase 3, multicenter, randomized, double-blind, parallel group study designed to describe the benefits and potential risks of a new treatment strategy using a fixed dose of darbepoetin alfa in subjects with CKD and not on dialysis. Anemic subjects without recent use of an erythropoiesis stimulating agent (ESA) will be randomly allocated 1:1 to treatment with a fixed dose of darbepoetin alfa or to treatment with darbepoetin alfa using a Hb-based titration strategy, which has been the conventional dosing strategy. In the Hb-based titration group, darbepoetin alfa doses will be titrated to maintain Hb ≥ 10.0 g/dL. This study aims to estimate the incidence of RBC transfusions (administered as deemed clinically necessary) in each group and the difference in incidence of RBC transfusions between the 2 groups. In addition, multiple aspects, such as cumulative darbepoetin alfa dose, total number of units of transfusions, Hb concentration, Hb-related parameters (eg, Hb variability, excursions, rate of change), and adverse (eg, cardiovascular) events, will also be considered in order to determine a preferred dosing regimen. Treatment group, darbepoetin alfa doses, and protocol specified Hb concentrations will be blinded to the investigator, subjects and study team. Subjects will be followed for approximately 2 years from the date of randomization.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical history of advanced CKD not on dialysis with at least 1 historic estimated glomerular filtration rate (eGFR) < 45.0 mL/mi)/1.73 m2 at least 12 weeks prior to screening
* Not currently receiving dialysis with an eGFR < 45.0 mL/min/1.73m2, per the central laboratory during screening
* Chronic anemia due to renal failure
* Two Hb concentrations < 10.0 g/dL, at least 2 weeks apart during screening using the modified Hb point of care (POC) device
* Iron replete, defined as a transferrin saturation (TSAT) ≥ 20% and a ferritin ≥ 100 ng/mL, per the central laboratory during screening
* Vitamin B12 and folate replete, defined as a vitamin B12 level > 180 pg/mL and a folate concentration > 7 nmol/L, per the central laboratory during screening
* Clinically stable in the opinion of the investigator
* Subject has provided written informed consent

Key Exclusion Criteria:

* Systemic hematologic disease (eg, sickle cell anemia, myelodysplastic syndrome, hematologic malignancy)
* Current or prior malignancy within 5 years of screening, with the exception of non-melanoma skin cancers and cervical intraepithelial neoplasia
* Treatment for any malignancy (eg, radiation, chemotherapy, hormone therapy, or biologics) within 5 years of screening, with the exception of locally excised non-melanoma skin cancer or cervical intraepithelial neoplasia
* Female subject not willing to use highly effective methods of birth control during treatment and for 4 weeks after the end of treatment
* Subject is pregnant or breast feeding, or might become pregnant during the study or within 4 weeks after the end of treatment
* Currently receiving intravenous (IV) antibiotics for treatment of an active infection
* Known Human Immunodeficiency Virus (HIV) positive
* Currently receiving systemic immunosuppressive therapy with the exception of prednis(ol)one ≤ 10 mg per day (or the steroid equivalent)
* History of any organ transplant
* Currently enrolled in another interventional study (eg, studies which require medical device use or drug therapy or with protocol required procedures), or less than 4 weeks since ending another interventional study(s) or receiving investigational agent(s)
* Known neutralizing anti-erythropoietic protein antibodies
* Known sensitivity to any of the products to be administered during dosing
* Previously enrolled in this study
* Not expected to be available for protocol required study visits or procedures to the best of the subject and investigator's knowledge
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with all required study procedures
* Occurrence of stroke or myocardial infarction (MI) within 24 weeks of screening
* Receipt of RBC transfusion within 8 weeks of screening
* Occurrence of seizure, clinically relevant active bleeding (eg, gastrointestinal [GI] bleed) or any hospitalization within 8 weeks of screening
* Receipt of any IV iron therapy within 4 weeks of screening
* Changes in oral iron therapy within 4 weeks of screening
* Receipt of ESA therapy within 4 weeks of screening
* Diagnosis or treatment of malignancy, with the exception of non-melanoma skin cancers and cervical intraepithelial neoplasia during screening
* Receipt of ESA therapy, RBC transfusions, IV iron therapy during screening
* Changes in oral iron therapy during screening
* Occurrence of stroke, MI, seizure, clinically relevant active bleeding (eg, GI bleed), any hospitalization or outpatient surgery during screening
* Uncontrolled hypertension during screening. Defined in this study, as a mean systolic blood pressure > 140 mmHg at both screening visits, or a mean systolic blood pressure >/= 160 mmHg at any screening visit, or a mean diastolic blood pressure >/= 90 mmHg at any screening visit.
* Expected or scheduled change in oral iron therapy or receipt of IV iron therapy within 4 weeks after randomization
* Expected or scheduled receipt of a RBC transfusion within 8 weeks after randomization
* Expected or scheduled organ transplant within 24 weeks after randomization
* Expected or scheduled initiation of dialysis within 24 weeks after randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (205):
- United States (201):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Goodyear, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Bell Gardens, California
  - Research Site, Beverly Hills, California
  - Research Site, Cerritos, California
  - Research Site, Chula Vista, California
  - Research Site, Cudahy, California
  - Research Site, El Centro, California
  - Research Site, Fountain Valley, California
  - Research Site, Fullerton, California
  - Research Site, Garden Grove, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, Huntington Beach, California
  - Research Site, Inglewood, California
  - Research Site, La Jolla, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Lakewood, California
  - Research Site, Lancaster, California
  - Research Site, Lomita, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Mission Hills, California
  - Research Site, Modesto, California
  - Research Site, Northridge, California
  - Research Site, Orange, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Dimas, California
  - Research Site, Whittier, California
  - Research Site, Yuba City, California
  - Research Site, Arvada, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Middlebury, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, North Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Hudson, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Summerfield, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Columbus, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Natchitoches, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Ruston, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Rockport, Maine
  - Research Site, Bethesda, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Framingham, Massachusetts
  - Research Site, Plymouth, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Southgate, Michigan
  - Research Site, Columbus, Mississippi
  - Research Site, Gulfport, Mississippi
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, North Platte, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Eatontown, New Jersey
  - Research Site, Livingston, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Flushing, New York
  - Research Site, Great Neck, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Orchard Park, New York
  - Research Site, Rochester, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Grand Forks, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Poland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Willoughby Hills, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Roseburg, Oregon
  - Research Site, Beaver, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Columbia, Tennessee
  - Research Site, Dyersburg, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, Edinburg, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Frisco, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Lufkin, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Mechanicsville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Silverdale, Washington
  - Research Site, Bluefield, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Puerto Rico (4):
  - Research Site, Caguas
  - Research Site, Ponce
  - Research Site, Rio Piedras
  - Research Site, San Juan

REFERENCES:
- [Background] Toto R, Petersen J, Berns JS, Lewis EF, Tran Q, Weir MR. A Randomized Trial of Strategies Using Darbepoetin Alfa To Avoid Transfusions in CKD. J Am Soc Nephrol. 2021 Feb;32(2):469-478. doi: 10.1681/ASN.2020050556. Epub 2020 Dec 7. PMID 33288629
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Anemic participants with chronic kidney disease and not on dialysis (CKD-ND) were enrolled at 126 study centers in the United States, from 30 July 2012 to 19 October 2017. The on-study duration was approximately 2 years, comprising of a 2- to 4-week screening period, a 96-week treatment period and a 4-week follow up period.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to 1 of 2 darbepoetin alfa dosing strategies (hemoglobin [Hb]-based titration group or fixed dose group). Randomization was stratified by red blood cell (RBC) transfusion received within 12 months prior to randomization (yes/no) and site practice setting (nephrology/non-nephrology).
Groups:
- Hb-Based Titration Group: Participants received darbepoetin alfa as a subcutaneous (SC) injection once every 4 weeks (Q4W) for up to 96 weeks. The dose of darbepoetin alfa was titrated based on the Hb concentration on the date of the visit, the corresponding Hb rate of rise (ROR), and the previously assigned dose. Doses were reduced if Hb exceeded 10.5 grams/deciliter (g/dL) or Hb ROR exceeded 1.0 g/dL/4W. When darbepoetin alfa therapy was withheld per the dosing algorithm, placebo was administered. The starting dose of darbepoetin alfa was 0.45 micrograms/kilogram (mcg/kg) and the protocol specified doses ranged from 10 to 300 mcg.
- Fixed Dose Group: Participants received darbepoetin alfa as a SC injection Q4W at the same dose as assigned at the time of randomization for the duration of the 96-week treatment period. There was 1 exception to the fixed dose strategy: if the Hb was > 12.0 g/dL, darbepoetin alfa therapy was withheld and placebo administered. Once the Hb fell to < 10.0 g/dL, darbepoetin alfa therapy resumed at the same dose. The starting dose of darbepoetin alfa was 0.45 mcg/kg and the protocol specified doses ranged from 10 to 300 mcg.
Period: Overall Study
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Started | 377 | 379
Received Investigational Product | 377 | 377
Completed | 232 | 226
Not Completed | 145 | 153
Not completed — Death | 36 | 39
Not completed — Lost to Follow-up | 28 | 23
Not completed — Decision by sponsor | 5 | 7
Not completed — Withdrawal by Subject | 76 | 84

BASELINE CHARACTERISTICS:
Groups:
- Hb-Based Titration Group: Participants received darbepoetin alfa as a SC injection, Q4W for up to 96 weeks. The dose of darbepoetin alfa was titrated based on the Hb concentration on the date of the visit, the corresponding Hb ROR, and the previously assigned dose. Doses were reduced if Hb exceeded 10.5 g/dL or Hb ROR exceeded 1.0 g/dL/4W. When darbepoetin alfa therapy was withheld per the dosing algorithm, placebo was administered. The starting dose of darbepoetin alfa was 0.45 mcg/kg and the protocol specified doses ranged from 10 to 300 mcg.
- Total: Total of all reporting groups
Arm/Group | Hb-Based Titration Group | Fixed Dose Group | Total
Number analyzed (Participants) | 377 | 379 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (13.5) | 69.5 (13.1) | 69.4 (13.3)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 129 | 134 | 263
  65 - 74 years | 97 | 96 | 193
  75 - 84 years | 105 | 97 | 202
  >=85 years | 46 | 52 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 218 | 441
  Male | 154 | 161 | 315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 92 | 95 | 187
  Not Hispanic or Latino | 285 | 284 | 569
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 25 | 21 | 46
  Black or African American | 125 | 134 | 259
  Native Hawaiian or Other Pacific Islander | 5 | 4 | 9
  White | 220 | 215 | 435
  Mixed race/Other | 1 | 5 | 6
Previous RBC transfusions [Count of Participants; unit: Participants]
  Yes | 145 | 140 | 285
  No | 232 | 239 | 471

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Receipt of 1 or More RBC Transfusions
Description: The percentage of participants receiving at least 1 RBC transfusion during the evaluation period was recorded for each treatment group. The evaluation period began from the date of randomization, and participants were censored at the last dose of investigational product plus 3 months or end of study, whichever was earlier (on-treatment approach).
Time Frame: From randomization until the end of study, up to week 101.
Population: The full analysis set included all randomized participants who received at least 1 dose of investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Number analyzed (Participants) | 377 | 377
Percentage of Participants | 24.40 [20.07 to 28.74] | 24.14 [19.82 to 28.46]
Statistical Analysis 1: Comparison: Hb-Based Titration Group vs Fixed Dose Group; Test type: Other; Treatment Difference = -0.27, 95% CI 2-sided [-6.39 to 5.85] — Difference is fixed dose - titration
Statistical Analysis 2: Comparison: Hb-Based Titration Group vs Fixed Dose Group; Test type: Other; Cochran-Mantel-Haenszel; Stratified by RBC transfusion received within 12 months prior to randomization (yes/no) and site practice setting (nephrology/non-nephrology); Risk Ratio (RR) = 0.998, 95% CI 2-sided [0.776 to 1.285] — A risk ratio < 1.0 indicates a lower event rate for the fixed dose group relative to Hb-based titration group

2. Secondary Outcome: Mean Number of Units of RBC Transfused
Description: The total number of units of RBC transfused per participant during the evaluation period was recorded for each treatment group. The evaluation period began from the date of randomization, and participants were censored at the last dose of investigational product plus 3 months or end of study, whichever was earlier (on-treatment approach). The mean total number of RBC units transfused per participant is presented.
Time Frame: From randomization until the end of study, up to week 101.
Population: The full analysis set included all randomized participants who received at least 1 dose of investigational product.
Measure: Mean (95% Confidence Interval); unit: Units of transfused RBC
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Number analyzed (Participants) | 377 | 377
Units of transfused RBC | 0.71 [0.53 to 0.89] | 0.87 [0.65 to 1.10]
Statistical Analysis 1: Comparison: Hb-Based Titration Group vs Fixed Dose Group; Test type: Other — Stratified by RBC transfusion received within 12 months prior to randomization (yes/no) and site practice setting (nephrology/non-nephrology) and accounting for participant exposure time; Negative binomial regression model; Least Squares Mean (LSM) Ratio = 1.28, 95% CI 2-sided [0.81 to 2.05] — Least Squares Mean (LSM) ratio is fixed dose relative to titration

3. Secondary Outcome: Time to First RBC Transfusion
Description: Time to first RBC transfusion during the evaluation period was recorded for each treatment group. The evaluation period began from the date of randomization, and participants were censored at the last dose of investigational product plus 3 months or end of study, whichever was earlier (on-treatment approach). The time to first RBC transfusion is presented using Kaplan-Meier (KM) estimates at 6, 12, 18, and 24 months.
Time Frame: From randomization until the end of study, up to week 101.
Population: The full analysis set included all randomized participants who received at least 1 dose of investigational product.
Measure: Number; unit: Months
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Number analyzed (Participants) | 377 | 377
Months
  KM estimates at month 6 | 0.115 | 0.136
  KM estimates at month 12 | 0.192 | 0.204
  KM estimates at month 18 | 0.261 | 0.246
  KM estimates at month 24 | 0.297 | 0.289
Statistical Analysis 1: Comparison: Hb-Based Titration Group vs Fixed Dose Group; Test type: Other; Cox Proportional Hazard Model; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.76 to 1.35] — Hazard ratio is fixed dose relative to titration

4. Secondary Outcome: Mean Achieved Hb Concentration While Receiving Investigational Product
Description: Average achieved Hb concentration while receiving investigational product was recorded as mean Hb using the area under the curve (AUC) method for each treatment group. The AUC of Hb was calculated according to the trapezoidal method, standardized as daily AUC. Participants with available Hb values from study day 85 (week 13) to the last dose date were included in the calculation.
Time Frame: From week 13 until the end of study, up to week 101.
Population: The full analysis set included all randomized participants who received at least 1 dose of investigational product.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Number analyzed (Participants) | 377 | 377
g/dL | 9.71 (0.04) | 9.41 (0.05)
Statistical Analysis 1: Comparison: Hb-Based Titration Group vs Fixed Dose Group; Test type: Other; Hodges-Lehmann estimate; Median of the difference = -0.34, 95% CI 2-sided [-0.46 to -0.22] — Difference is fixed dose - titration; The 2-sided 95% confidence intervals were obtained using a non-parametric Wilcoxon rank-sum statistic

5. Secondary Outcome: Geometric Mean Cumulative Dose of Darbepoetin Alfa Per 4 Weeks
Description: Cumulative doses of darbepoetin alfa adjusted for investigation product exposure time (e.g. mean cumulative darbepoetin alfa dose per 4 weeks) were calculated for each treatment group using the total cumulative dose during the study divided by total number of weeks dosed then multiplied by 4. The geometric mean cumulative dose is presented.
Time Frame: From randomization until the end of study, up to week 101.
Population: The full analysis set included all randomized participants who received at least 1 dose of investigational product.
Measure: Geometric Mean (Standard Error); unit: mcg
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
Number analyzed (Participants) | 377 | 377
mcg | 50.7 (2.7) | 30.8 (1.2)
Statistical Analysis 1: Comparison: Hb-Based Titration Group; Test type: Other; Hodges-Lehmann estimate; Median of the difference = -22.1, 95% CI 2-sided [-26.1 to -18.1] — Difference is fixed dose - titration; The 2-sided 95% confidence intervals were obtained using a non-parametric Wilcoxon rank-sum statistic

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were collected from randomization on study day 1 until 4 weeks after final dose of investigational product (up to 101 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Hb-Based Titration Group | Fixed Dose Group
All-Cause Mortality (participants affected / at risk) | 38/377 | 38/377
Serious Adverse Events (participants affected / at risk) | 190/377 | 175/377
Other Adverse Events (participants affected / at risk) | 292/377 | 300/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hb-Based Titration Group (N=377) | Fixed Dose Group (N=377)
Anaemia (Blood and lymphatic system disorders) | 24 | 29
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Hyperprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 5
Angina pectoris (Cardiac disorders) | 3 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 1
Cardiac arrest (Cardiac disorders) | 3 | 3
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 11 | 7
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 28 | 17
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 3
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 3
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 4 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 3
Death (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 2 | 2
Hypothermia (General disorders) | 0 | 2
Influenza like illness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 6 | 1
Oedema peripheral (General disorders) | 4 | 2
Peripheral swelling (General disorders) | 1 | 0
Pneumatosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Abscess limb (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 3 | 5
Cholecystitis infective (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Emphysematous pyelonephritis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 1 | 0
Mycobacterium kansasii infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 3
Osteomyelitis acute (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 15 | 18
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyuria (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 3
Septic shock (Infections and infestations) | 1 | 2
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal urinary tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 9 | 11
Urinary tract infection bacterial (Infections and infestations) | 2 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 10 | 2
Femur fracture (Injury, poisoning and procedural complications) | 4 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Acid base balance abnormal (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
ECG signs of myocardial ischaemia (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 10 | 5
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Dysarthria (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 5 | 6
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Device leakage (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Drug abuse (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 34 | 24
Azotaemia (Renal and urinary disorders) | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 5 | 4
End stage renal disease (Renal and urinary disorders) | 12 | 6
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 7 | 5
Renal impairment (Renal and urinary disorders) | 2 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Dialysis (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Diastolic hypertension (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 6 | 3
Hypertensive crisis (Vascular disorders) | 4 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 4
Intermittent claudication (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hb-Based Titration Group (N=377) | Fixed Dose Group (N=377)
Anaemia (Blood and lymphatic system disorders) | 19 | 36
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 3 | 5
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve sclerosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 5 | 4
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 6
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 5
Cardiomegaly (Cardiac disorders) | 2 | 7
Cardiomyopathy (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 2 | 0
Dilatation atrial (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dilatation (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve calcification (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 3
Pulmonary valve incompetence (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 2
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Vascular malformation (Congenital, familial and genetic disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 4 | 5
Adrenal mass (Endocrine disorders) | 1 | 0
Hyperadrenalism (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 2 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 3 | 3
Hypothyroidism (Endocrine disorders) | 3 | 5
Secondary hyperthyroidism (Endocrine disorders) | 1 | 0
Astigmatism (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 6 | 4
Cataract cortical (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Diabetic retinal oedema (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 2
Dry eye (Eye disorders) | 1 | 3
Eye allergy (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 1 | 2
Hypermetropia (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 0 | 1
Presbyopia (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 11 | 17
Dental caries (Gastrointestinal disorders) | 1 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 19
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 7
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 8
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 3
Hiatus hernia (Gastrointestinal disorders) | 2 | 4
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 2
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 27 | 22
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 4
Toothache (Gastrointestinal disorders) | 3 | 4
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 17 | 12
Asthenia (General disorders) | 17 | 15
Chest discomfort (General disorders) | 3 | 0
Chest pain (General disorders) | 8 | 10
Chills (General disorders) | 5 | 2
Cyst (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Fatigue (General disorders) | 17 | 21
Feeling cold (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 1
Influenza like illness (General disorders) | 3 | 3
Injection site oedema (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 2
Oedema (General disorders) | 17 | 18
Oedema peripheral (General disorders) | 35 | 29
Pain (General disorders) | 5 | 4
Peripheral swelling (General disorders) | 8 | 9
Polyp (General disorders) | 2 | 0
Pyrexia (General disorders) | 6 | 4
Sluggishness (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 0 | 1
Thirst (General disorders) | 2 | 0
Vaccination site bruising (General disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 2
Seasonal allergy (Immune system disorders) | 2 | 3
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 1
Abscess neck (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 5 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 1
Blister infected (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 19 | 15
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 8 | 9
Chikungunya virus infection (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Coccidioidomycosis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 2
Conjunctivitis bacterial (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 2 | 4
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Ear infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 1
Fungal skin infection (Infections and infestations) | 4 | 2
Furuncle (Infections and infestations) | 1 | 2
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 3
Genital candidiasis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 2
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 6 | 5
Infected cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 5
Laryngitis (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 16
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 2 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 2 | 0
Periorbital abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyoderma (Infections and infestations) | 0 | 1
Pyuria (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sebaceous gland infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 6 | 6
Sinusitis bacterial (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 2 | 4
Tooth infection (Infections and infestations) | 1 | 3
Trichomoniasis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 19 | 26
Urinary tract infection (Infections and infestations) | 38 | 35
Urinary tract infection bacterial (Infections and infestations) | 1 | 3
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 1
Viral rhinitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 8 | 16
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 26 | 22
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 6 | 8
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 2
Limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 4
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 3 | 3
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 3
Skin injury (Injury, poisoning and procedural complications) | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Tooth avulsion (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 4 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood iron decreased (Investigations) | 1 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0
Blood phosphorus increased (Investigations) | 2 | 0
Blood potassium abnormal (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Blood pressure abnormal (Investigations) | 1 | 0
Blood pressure diastolic (Investigations) | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 24 | 16
Blood pressure systolic increased (Investigations) | 1 | 2
Carbon dioxide decreased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 1 | 0
Computerised tomogram abnormal (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Endoscopy gastrointestinal normal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Protein total increased (Investigations) | 0 | 1
Serum ferritin decreased (Investigations) | 1 | 0
Thyroid function test abnormal (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Tuberculin test positive (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 3 | 3
Weight increased (Investigations) | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 13
Dehydration (Metabolism and nutrition disorders) | 6 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 5 | 6
Gout (Metabolism and nutrition disorders) | 12 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 3
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 18 | 39
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 7
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Iron deficiency (Metabolism and nutrition disorders) | 4 | 6
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 13
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 22
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
CREST syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 12
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 3 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 13 | 28
Dizziness postural (Nervous system disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 14
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 6
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 3
Seizure (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 7 | 3
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 5 | 6
Hallucination (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 6 | 11
Mental status changes (Psychiatric disorders) | 2 | 5
Paranoia (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 10 | 6
Anuria (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 3 | 0
Bladder mass (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 9 | 14
Dysuria (Renal and urinary disorders) | 4 | 5
End stage renal disease (Renal and urinary disorders) | 4 | 5
Haematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Polyuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2
Renal atrophy (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 2 | 3
Renal mass (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 3
Breast mass (Reproductive system and breast disorders) | 1 | 0
Breast ulceration (Reproductive system and breast disorders) | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 2
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 2
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 6
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 10
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 6
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 2
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 2 | 3
Catheter placement (Surgical and medical procedures) | 0 | 2
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Nephrostomy (Surgical and medical procedures) | 1 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0
Toe operation (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 3 | 0
Angiopathy (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Diastolic hypotension (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 46 | 40
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 22
Intermittent claudication (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2013-12-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT01652872/Prot_000.pdf
  • Statistical Analysis Plan (2012-05-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT01652872/SAP_001.pdf